CLINICAL TRIAL: NCT05809024
Title: Select the Appropriate Population for Adding CDK4/6i to Neoadjuvant Endocrine Therapy in High Risk Early HR+/HER2-breast Cancer Based on Molecular Marker
Brief Title: Select the Appropriate Population for Adding CDK4/6i to Neoadjuvant Endocrine Therapy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yongsheng Wang (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yongsheng Wang, Director of breast cancer center, Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-023
Record Dates: First submitted 2023-03-29; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Locally Advanced Breast Cancer; Hormone Receptor Positive，HER2-negative Breast Cancer
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single Arm (Experimental): Hormone receptor positive,HER2 negative participants will receive letrozole as neoadjuvant endocrine therapy，if ki67 was higher than 10% after two weeks,CDK4/6 Inhibitor was added.
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: letrozole — Hormone receptor positive,HER2 negative participants will receive letrozole as neoadjuvant endocrine therapy，if don't work, CDK4/6 Inhibitor was added.
  Other Names: CDK4/6 Inhibitor

SUMMARY:
Select the appropriate population for adding CDK4/6 inhibitors therapy in high risk early HR+/HER2-breast cancer based on molecular detection

ELIGIBILITY:
Inclusion Criteria:

1. Newly treated female patients, ≥18 and ≤75 years;
2. ECOG score 0-1;
3. Breast cancer following:

   Histologically confirmed invasive breast cancer with primary tumor diameter >2 cm by standard evaluation methods.Tumor stage: cT2-cT4/cN0-cN3/cM0 (clinical phase II and III)
4. HR+/HER2- breast cancer confirmed by pathological examination, defined as: primary HR+/HER2- breast cancer performed by the pathology department of the Central Hospital;
5. Get hormone receptor status (ER and PR);
6. Major organ function following:

   Complete blood count: Neutrophil (ANC) ≥ 1.5×109/L; Platelet count (PLT) ≥ 90×109/L; hemoglobin (Hb) ≥90 g/L; Blood Biochemistry: Total bilirubin (TBIL) ≤ 2.5×ULN; Alanine aminotransferase (ALT) ≤ 1.5×ULN; Aspartate aminotransferase (AST) ≤ 1.5×ULN; Alkaline phosphatase ≤ 2.5×ULN; Urea nitrogen (BUN) ≤ 1.5×ULN; Creatinine (Cr) ≤ 1.5×ULN; Twelve-lead electrocardiogram: Fridericia corrected QT Interval (QTcF) woman < 470 ms (QTcF=QT/(RR^1/3));
7. Woman who are not menopausal or have not been surgically sterilized agree to abstain from sex or use effective contraceptive methods for at least the duration of the study treatment and for 7 months after the last dosing;
8. Volunteer to participate in the study, sign informed consent, have good compliance and be willing to cooperate with follow-up.

Exclusion Criteria:

1. IV stage breast cancer or metastatic breast cancer;
2. Inflammatory breast cancer;
3. Any previous malignant tumor or previous anti-tumor therapy or radiotherapy were not allowed, excluding cured cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma;
4. Participate in other clinical trials;
5. Patients were not allowed who had undergone major non-breast cancer related surgery within 4 weeks prior to randomization or had not fully recovered from such surgery;
6. Patients were not allowed who had received blood transfusion or colony stimulating factor treatment within 2 weeks before randomization;
7. Patients were not allowed who allergic to drug components;
8. Patients were not allowed who had a history of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
9. Patients have heart disease were not allowed including: (1) angina pectoris; (2) medically treatable or clinically significant arrhythmias; (3) myocardial infarction; (4) heart failure; (5) any other heart disease that the investigator has determined is not suitable for participation in the study;
10. Pregnant and lactating women, fertile women who tested positive for baseline pregnancy tests, or fertile women who were unwilling to take effective contraceptive measures during the test period were not allowed;
11. Patients have concomitant diseases that endanger patient safety or influence the completion of the study were not allowed (including but not limited to hypertension, severe diabetes, active infection, thyroid disease, etc.);
12. Patients were not allowed who with inability to swallow, chronic diarrhea and intestinal obstruction, accompany multiple factors affecting the administration and absorption of medicines;
13. Any other circumstances in which the investigator considers the patients unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
ki67 index | Up to approximately 2 weeks
  Independent review committee (IRC) evaluates the Ki67 index after treatment. Ki67 index using the definition of HE stained breast cancer samples after neoadjuvant therapy and surgery. (Defined by the American Joint Committee onCancer, AJCC).

SECONDARY OUTCOMES:
Objective Overall Response Rate | Up to approximately 7 weeks
  Defined as the proportion of subjects who achieved CR or PR as optimal tumor response during neoadjuvant therapy. Objective response rates will be assessed according to the RECIST v1.1 for the evaluation of efficacy in solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: yongsheng wang, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Breast Cancer Center, Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No